CLINICAL TRIAL: NCT04817813
Title: LIBREAST STUDY: Long-term Outcomes After Breast Cancer Liver Metastasis Surgery: an European, Retrospective, Snapshot Study
Brief Title: Long-term Outcomes After Breast Cancer Liver Metastasis Surgery: an European, Retrospective, Snapshot Study
Acronym: LIBREAST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Miguel Servet (Other)
Collaborators: Spanish Association of Surgeons (AEC) (Other)
Responsible Party: Principal Investigator, Mario Serradilla, MD, FACS, Principal Investigator, Hospital Miguel Servet
Other Study IDs: PI20/596
Record Dates: First submitted 2021-02-05; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer; Liver Metastases; Surgery
Keywords: Breast cancer; Liver metastases; Hepatic surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer ranks as the top leading malignant tumors among females, and also accounts for the most common cause of tumor related mortality in females worldwide. Approximately, 20-30% of breast cancer cases develop metastasis, while 50% of patients will suffer from breast cancer liver metastasis. The proper indication for surgical treatment of breast cancer liver metastasis is still a matter of discussion. Surgery is becoming more practical and effective than conservative treatment in improving the outcomes of patients with breast cancer liver metastasis and liver metastasis surgery is included in an onco- surgical strategy.

DETAILED DESCRIPTION:
Breast cancer ranks as the top leading malignant tumors among females, and also accounts for the most common cause of tumor related mortality in female's worldwide . Approximately, 20-30% of breast cancer (BC) cases develop metastasis, while 50% of patients will suffer from breast cancer liver metastases (BCLM) . The presence of liver metastasis has markedly worsened the prognosis of patients, and the median survival was reported to be 3.8-29 months.

Metastatic breast cancer is considered to be a disseminated disease and many oncologists remain reluctant to include surgery within the multimodal treatment strategy of these patients . Although systemic treatments can achieve approximately 60% of responses in breast cancer recurrence, long-term survival is exceptional only with medical treatment . Without liver resection, the average survival reported after the first onset of liver metastases is distributed over a range from 1 to 15 months. Surgery is becoming more functional and effective than conservative treatment in improving the poor outcomes of patients with BCLM . However, there is no generally acknowledged set of standards for identifying candidates who will benefit from surgery. The proper indication for surgical treatment is still a matter of discussion; surgical resection should be assessed when the following premises are met: low surgical risk, low metastasis number, complete macroscopic liver removal, absence of proven extrahepatic disease by positron emission tomography and computed tomography, objective response to chemotherapy before surgery, and long disease-free interval. Breast cancer liver metastasis surgery (BCLMS) is included in an onco-surgical strategy.

Most of the published series of patients with liver metastases of breast cancer who have undergone surgery come from a single center or few centers and there are hardly any long-term results, so we consider necessary to carry out a multicenter review of patients who underwent surgery in high volume centers across Europe belonging to the European-African Hepato-Pancreato-Biliary Association (E-AHPBA) to asses survival and disease-free survival and to determine which patients may benefit from surgery.

This retrospective multicenter cohort study in centers performing BCLMS aims to provide an assessment of the outcomes across E-AHPBA centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 year old.
* Scheduled surgery for breast cancer liver metastases between January 1st 2010 and December 31st 2015
* American Society of Anesthesiologists (ASA) score I-III.
* They have signed the informed consent.

Exclusion Criteria:

* Patients under 18 year old.
* ASA ≥ IV.
* Urgent surgery.
* Patients who have not signed the informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients operated on in the participating European centers with breast cancer liver metastases during the study period (between January 1st 2010 and December 31st 2015) and that meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Survival and disease-free survival at 1st year. | 1 year.
  Disease-free time and survival at 1st year.
Survival and disease-free survival at 3th year. | 3 years.
  Disease-free time and survival at 3th year.
Survival and disease-free survival at 5th year. | 5 years.
  Disease-free time and survival at 5th year.

SECONDARY OUTCOMES:
Preoperative details-Tumor TNM | 5 years.
  Stage
Preoperative details- Dysplasia grade | 5 years.
  Low-Moderate- High
Preoperative details- Tumor subtypes | 5 years.
  Yes/No of Luminal A/Luminal B/ HER2+/Triple negative-basal like
Preoperative details- Location of breast cancer | 5 years.
  Breast Quadrant
Preoperative details- Segment location | 5 years.
  Segment 1 to 8
Preoperative details- Number of liver metastasis | 5 years.
  Number
Intra-operative events | Surgery date.
  Satava's Classification
Nº metastasis intraoperatively | Surgery date.
  Number
Post-operative curse- Re-hospitalization cause | 30 days.
  Cause of re-hospitalization
Post-operative curse- Complications | 30 days.
  Clavien- Dindo Classification
Post-operative curse- ICU admission length of stay | 30 days.
  Days
Histopathological details- Ki67 | 30 days.
  Percent
Histopathological details- Resection status | 30 days.
  R0-R1-R2
Histopathological details- Nº of lesions | 30 days.
  Number
Follow up- Adjuvant systemic treatment | 5 years.
  Yes/No of Chemotherapy, Hormonetherapy, AntiHER2Therapy, Antiangiogenics
Follow up- Liver metastasis relapse | 5 years.
  Location of relapse
Follow up- Date of death | 5 years.
  Date

CONTACTS AND LOCATIONS:
Overall Officials: Mario Serradilla Martín, MD FACS, Principal Investigator — Zaragoza, Spain. Miguel Servet University Hospital
Locations (1):
- Mario Serradilla Martín, Zaragoza, Spain

REFERENCES:
- [Result] He X, Zhang Q, Feng Y, Li Z, Pan Q, Zhao Y, Zhu W, Zhang N, Zhou J, Wang L, Wang M, Liu Z, Zhu H, Shao Z, Wang L. Resection of liver metastases from breast cancer: a multicentre analysis. Clin Transl Oncol. 2020 Apr;22(4):512-521. doi: 10.1007/s12094-019-02155-2. Epub 2019 Jun 22. PMID 31230220
- [Result] Chen QF, Huang T, Shen L, Wu P, Huang ZL, Li W. Prognostic factors and survival according to tumor subtype in newly diagnosed breast cancer with liver metastases: A competing risk analysis. Mol Clin Oncol. 2019 Sep;11(3):259-269. doi: 10.3892/mco.2019.1890. Epub 2019 Jul 1. PMID 31396386
- [Result] Sadot E, Lee SY, Sofocleous CT, Solomon SB, Gonen M, Kingham TP, Allen PJ, DeMatteo RP, Jarnagin WR, Hudis CA, D'Angelica MI. Hepatic Resection or Ablation for Isolated Breast Cancer Liver Metastasis: A Case-control Study With Comparison to Medically Treated Patients. Ann Surg. 2016 Jul;264(1):147-154. doi: 10.1097/SLA.0000000000001371. PMID 26445472
- [Result] Margonis GA, Buettner S, Sasaki K, Kim Y, Ratti F, Russolillo N, Ferrero A, Berger N, Gamblin TC, Poultsides G, Tran T, Postlewait LM, Maithel S, Michaels AD, Bauer TW, Marques H, Barroso E, Aldrighetti L, Pawlik TM. The role of liver-directed surgery in patients with hepatic metastasis from primary breast cancer: a multi-institutional analysis. HPB (Oxford). 2016 Aug;18(8):700-5. doi: 10.1016/j.hpb.2016.05.014. Epub 2016 Jun 29. PMID 27485066
- [Result] Treska V, Cerna M, Kydlicek T, Treskova I. Prognostic factors of breast cancer liver metastasis surgery. Arch Med Sci. 2015 Jun 19;11(3):683-5. doi: 10.5114/aoms.2015.52376. No abstract available. PMID 26170865
- [Result] Diaz R, Santaballa A, Munarriz B, Calderero V. Hepatic resection in breast cancer metastases: should it be considered standard treatment? Breast. 2004 Jun;13(3):254-8. doi: 10.1016/j.breast.2003.11.001. PMID 15177433
- [Result] Ramia JM, Villar J, Villegas T, Muffak K, Garrote D, Ferron JA. [Surgical treatment of liver metastases from breast cancer]. Cir Esp. 2005 Nov;78(5):318-22. doi: 10.1016/s0009-739x(05)70942-8. Spanish. PMID 16420849
- [Result] Figueras J, Gonzalez HD. [Surgical treatment of breast cancer liver metastasis. The great assignment awaiting Spanish hepatic surgery]. Cir Esp. 2008 Nov;84(5):239-40. doi: 10.1016/s0009-739x(08)75913-x. No abstract available. Spanish. PMID 19080906
- [Result] Roffman CE, Buchanan J, Allison GT. Charlson Comorbidities Index. J Physiother. 2016 Jul;62(3):171. doi: 10.1016/j.jphys.2016.05.008. Epub 2016 Jun 11. No abstract available. PMID 27298055
- [Result] Satava RM. Identification and reduction of surgical error using simulation. Minim Invasive Ther Allied Technol. 2005;14(4):257-61. doi: 10.1080/13645700500274112. PMID 16754172
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] The Royal College of Pathologists. Standards and Minimum Datasets for Reporting Cancers Minimum dataset for the histopathological reporting of pancreatic, ampulla of Vater and bile duct carcinoma. London R Coll Pathol. 2002.
- [Result] Rahbari NN, Garden OJ, Padbury R, Maddern G, Koch M, Hugh TJ, Fan ST, Nimura Y, Figueras J, Vauthey JN, Rees M, Adam R, Dematteo RP, Greig P, Usatoff V, Banting S, Nagino M, Capussotti L, Yokoyama Y, Brooke-Smith M, Crawford M, Christophi C, Makuuchi M, Buchler MW, Weitz J. Post-hepatectomy haemorrhage: a definition and grading by the International Study Group of Liver Surgery (ISGLS). HPB (Oxford). 2011 Aug;13(8):528-35. doi: 10.1111/j.1477-2574.2011.00319.x. Epub 2011 Jun 7. PMID 21762295
- [Result] Brooke-Smith M, Figueras J, Ullah S, Rees M, Vauthey JN, Hugh TJ, Garden OJ, Fan ST, Crawford M, Makuuchi M, Yokoyama Y, Buchler M, Weitz J, Padbury R. Prospective evaluation of the International Study Group for Liver Surgery definition of bile leak after a liver resection and the role of routine operative drainage: an international multicentre study. HPB (Oxford). 2015 Jan;17(1):46-51. doi: 10.1111/hpb.12322. Epub 2014 Jul 24. PMID 25059275
- [Result] Rahbari NN, Garden OJ, Padbury R, Brooke-Smith M, Crawford M, Adam R, Koch M, Makuuchi M, Dematteo RP, Christophi C, Banting S, Usatoff V, Nagino M, Maddern G, Hugh TJ, Vauthey JN, Greig P, Rees M, Yokoyama Y, Fan ST, Nimura Y, Figueras J, Capussotti L, Buchler MW, Weitz J. Posthepatectomy liver failure: a definition and grading by the International Study Group of Liver Surgery (ISGLS). Surgery. 2011 May;149(5):713-24. doi: 10.1016/j.surg.2010.10.001. Epub 2011 Jan 14. PMID 21236455
- [Derived] Cantalejo-Diaz M, Ramia JM, Alvarez-Busto I, Kokas B, Blanco-Fernandez G, Munoz-Forner E, Olah A, Montalva-Oron E, Lopez-Lopez V, Rotellar F, Eker H, Rijken A, Prieto-Calvo M, Romano F, Melgar P, Machairas N, Demirli Atici S, Castro-Santiago MJ, Lesurtel M, Skalski M, Bayhan H, Domingo-Del-Pozo C, Hahn O, de Armas-Conde N, Bauza-Collado M, Serradilla-Martin M; Scientific & Research Committee of the E-AHPBA. Long-term outcomes after breast cancer liver metastasis surgery: A European, retrospective, snapshot study (LIBREAST STUDY). Surg Oncol. 2024 Dec;57:102129. doi: 10.1016/j.suronc.2024.102129. Epub 2024 Sep 5. PMID 39243418